CLINICAL TRIAL: NCT06094855
Title: Effect of Cooling on Balance Performance in Persons With Multiple Sclerosis
Brief Title: Effect of Cooling on Balance Performance in Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: Hunter College of City University of New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0489-Hunter
Record Dates: First submitted 2023-09-25; First posted 2023-10-23 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons with Multiple sclerosis: Persons with a diagnosis of Multiple Sclerosis
  Interventions: Other: 20 minutes of biking on a stationary recumbent bicycle with and without a cooling vest

INTERVENTIONS:
Other: 20 minutes of biking on a stationary recumbent bicycle with and without a cooling vest — 2 bouts of 20 minutes of pedaling on a stationary recumbent bicycle, 1-2 weeks apart. Subjects will be cooled for one of the bouts and uncooled for the other.

SUMMARY:
The goal of this observational study to examine the effects of cooling on balance in persons with Multiple Sclerosis. Persons with Multiple Sclerosis frequently have problems with balance leading to falls and related injuries, as well as avoidance of activities that may challenge balance. Persons with Multiple Sclerosis are also well known to experience worsening of their symptoms when they become too warm, a condition known as thermosensitivity. This suggests that heat may worsen balance and increase falls risk in persons with Multiple Sclerosis. In this study we are examining the effects of wearing a cooling vest on balance performance in persons with MS. The main questions our study aims to answer are:

Question 1- Does wearing a cooling vest result in better balance performance in persons with MS when compared to a condition when they are not wearing the vest.

Participants will be given a balance test to assess their baseline balance performance. Following the test participants will be randomly assigned to either a cooled or an uncooled condition. In the cooled condition, participants will wear a commercially available cooling vest while pedaling for 20 minutes at their best comfortable pace on a recumbent stationary bicycle. Immediately following the 20 minutes of exercise the vest shall be removed and the balance test repeated. Subjects in the uncooled condition will perform the same task but without wearing the vest. One week later, participants will return and will perform the opposite of what they did the previous week; subjects who were in the cooled group will perform the 20 minute exercise test without the cooling vest and subjects who were uncooled will perform the test with a cooling vest. The same balance test will be performed before and after the exercise bout.The change in the balance scores between the 2 conditions will be compared.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effectiveness of cooling on balance performance on persons with MS(pwMS). Multiple studies have provided evidence that cooling can improve gait performance in MS; this will be the first study that examines the effect of cooling on balance. We hypothesize that persons with MS will have better balance performance when cooled, as opposed to a non-cooled condition. If our hypothesis is correct, it will suggest that physical therapists who work with pwMS can use cooling as a modality to improve balance. Outcomes will be shared via conference presentations through American Physical Therapy Association, Consortium of Multiple Sclerosis Centers, and publications in peer-reviewed journals. Results will also be shared with academic colleagues at other teaching centers.

Although cooling has been studied for its effects on gait in pwMS, our study will be the first to observe its effectiveness in improving balance. We are operationally defining improvement in balance by increase in score in the mini Balance Evaluation Systems Test, a valid and reliable tool for measuring balance and performance in MS. We are operationally defining cooling by the wearing of a commercially available cooling vest. Participants will be identified by contacting local area MS practices and support groups as well as posting our study on ClinicalTrials.gov. Consent will be obtained at the physical therapy department of Hunter College. Consent is obtained when the potential subject arrives prior to obtaining any demographic or subject characteristic information. As this is a randomized crossover trial, participants will be randomized into either a cooled or non-cooled condition. Following completion of experiencing one condition, they will then "cross over" and experience the other condition; subjects previously in the cooled group will cross over to the uncooled group and subjects in the uncooled group will crossover into the cooled group. Procedures will take place in the Physical Therapy department at Hunter College. Each subject will have to attend the Hunter College Physical Therapy department for 60-90 minutes, 2 times, 1-2 weeks apart. Prior to randomization, the following demographic and subject characteristic data will be collected: 1. Subject demographics and characteristics, 2. Multiple Sclerosis Impact Scale 29 (MSIS-29), 3. Fatigue Severity Scale, 4. Mini BESTest, 5. Activities-specific Balance Confidence Scale (ABC), This data will be collected to get a better description of the subject. Data will be collected on paper forms. There will not be interview/focus groups/survey questions.

Following collection of this data subjects will be randomized into either a cooled or uncooled condition via picking odd or even numbers out of a hat.

Subjects will then ride a stationary bicycle in order to induce fatigue. The protocol for the stationary bike ride is as follows:

Depending on randomization, subjects will ride the stationary bike either wearing the cooling vest (cooled condition) or not (uncooled condition). Immediately after the biking the subjects will repeat the Mini Balance Evaluation Systems Test. One week later, the subjects will return and repeat the balance testing and biking but in the opposite condition to what they were tested in previously.

ELIGIBILITY:
Inclusion Criteria: 1-Definitive diagnosis of Multiple Sclerosis 2-Capable of standing unassisted for at least 1 minute 3-ability to read and understand an informed consent 4- age 18-75

Exclusion Criteria:

1. Any orthopedic, cardiopulmonary, or non-MS neurologic complication that would interfere with balance because it is study on Multiple Sclerosis.
2. Under age 18 or over 75

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Community dwelling adults with Multiple Sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mini Balance Systems Evaluation Test | The test takes 15-20 minutes to administer. It will be administered 4 times; immediately before and immediately after the cooled cycling condition and immediately before before and immediately after the uncooled cycling condition.
  The MBT is a valid and reliable tool used to measure balance performance and falls risk in persons with MS.

SECONDARY OUTCOMES:
Visual Analog Scale of Fatigue | The test takes less than 1 minute to administer; It will be administered 4 times; immediately before and immediately after the cooled cycling condition and immediately before and immediately after the uncooled cycling condition.
  The Visual Analog Scale of Fatigue is used to measure subjective feelings of fatigue during a performance of a specific task.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Karpatkin, Dsc, Principal Investigator — Hunter College Physical therapy Department, City University of New York
Locations (1):
- Hunter College, Physical Therapy Department, City University of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No